CLINICAL TRIAL: NCT01453036
Title: Eradication of Helicobacter Pylori According to 23S rRNA Point Mutations Associated With Clarithromycin Resistance
Brief Title: Clarithromycin Resistant Tailored Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jin Il Kim (Other)
Collaborators: Korean College of Helicobacter and Upper Gastrointestinal Research (Other)
Responsible Party: Sponsor-Investigator, Jin Il Kim, professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUK
Record Dates: First submitted 2011-09-29; First posted 2011-10-17 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-07

CONDITIONS: Peptic Ulcer; Helicobacter Pylori Infection
Keywords: Peptic ulcer; Helicobacter pylori; Clarithromycin; 23S rRNA; Resistance
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional AOC group (Active Comparator): The investigators do not perform mutation test in the conventional group apply amoxicillin 1 g, bid , rabeprazole 20 mg bid, clarithromycin 500 mg bid during 1weeks
  Interventions: Procedure: UBT test & Gastroenterology with biopsy c silver stain
- Mutation test group (Active Comparator): Mutation test group is composed of two groups, clarithromycin group and metronidazole group Clarithromycin subgroup ; no point mutation at 23S rRNA apply clarithromycin 500 mg bid, amoxicillin 1 g bid, rabeprazole 20 mg bid during 1 week Metronidazole subgroup ; point mutation at 23S rRNA apply metronidazole 500 mg tid, amoxicillin 1 g bid, rabeprazole 20 mg bid during 1 week
  Interventions: Procedure: 23S rRNA point mutation test of Helicobacter pylori; Procedure: UBT test & Gastroenterology with biopsy c silver stain
- Conventional AOM group (Active Comparator): The investigators do not perform mutation test in the conventional group apply metronidazole 500 mg tid, amoxicillin 1 g bid, rabeprazole 20 mg bid during 1 week
  Interventions: Procedure: UBT test & Gastroenterology with biopsy c silver stain

INTERVENTIONS:
Procedure: 23S rRNA point mutation test of Helicobacter pylori — mutation test group>> Helicobacter pylori polymerase chain reaction kit by dual-priming oligonucleotide-based multiplex polymerase chain reaction system before eradication of Helicobacter pylori at mutation test groupConventional Conventional AOC group, Conventional AOM group >> no intervention
  Other Names: Seeplex ClaR-Helicobacter pylori polymerase chain reaction kit of Seegene Incorporated, Seoul, Korea
  Arms: Mutation test group
Procedure: UBT test & Gastroenterology with biopsy c silver stain — UBT test & Gastroenterology with biopsy c silver stain due to indentify H. pylori infection Conventional AOM group, Conventional AOC group, Mutation test group >> intervention

SUMMARY:
1. Back ground Antibiotics resistance of Helicobacter pylori, especially to clarithromycin is one of the main causes of failure of eradication. 23S rRNA point mutation of Helicobacter pylori is associated clarithromycin resistance
2. Hypothesis If the investigators check the 23S rRNA point mutation then choose treatment regimens containing a proton pump inhibitor and combination of two antibiotics (amoxicillin and clarithromycin or metronidazole), the investigators will eradicate Helicoabacter pylori more successfully
3. Material & methods The investigators enroll patients diagnosed with peptic ulcer, endoscopically. Helicobacter pylori is documented with Urea breath test or silver staining biopsy specimen or polymerase chain reaction of biopsy specimen. Check the 23S rRNA A2142G/A2143G point mutation by polymerase chain reaction. If there is mutation, the investigators consider as resistance to clarithromycin and choose the treatment regimen containing a proton pump inhibitor, amoxicillin, metronidazole. If there is no mutation, choose the treatment regimen containing a proton pump inhibitor, amoxicillin, clarithromycin. Verify Helicobacter pylori eradication by urea breath test. Compare eradication rate with conventional treatment,proton pump inhibitor, amoxicillin, clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 75 years old
* Peptic ulcer (gastric ulcer, duodenal ulcer)
* Helicobacter pylori positive

Exclusion Criteria:

* Major comorbidities
* Pregnancy
* History of Helicobacter pylori eradication
* History of gastric surgery or other cancers, except to endoscopic treatment due to gastric lesion

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jeong Lee, fellow, Principal Investigator — Yeouido St. Mary's Hospital, The Catholic University of Korea; Dae Young Cheung, professor, Principal Investigator — Yeouido St. Mary's Hospital, The Catholic University of Korea; Seong Su Kim, professor, Principal Investigator — The Catholic University of Korea; Byeong Ug Kim, Principal Investigator — The Catholic University of Korea; Tae Ho Kim, Principal Investigator — The Catholic University of Korea; Eun Jung Jeon, Principal Investigator — The Catholic University of Korea; Jung Hwan Oh, Professor, Principal Investigator — The Catholic University of Korea; Woo Chul Chung, professor, Principal Investigator — The Catholic University of Korea; Soo Heon Park, Principal Investigator — The Catholic University of Korea; Jea Kwang Kim, Principal Investigator — The Catholic University of Korea; Jin Il Kim, Study Chair — The Catholic University of Korea
Locations (1):
- Gastroenterology Clinic, Seoul, Yeouido-dong/Yeongdeungpo-gu, South Korea

REFERENCES:
- [Result] Cho DK, Park SY, Kee WJ, Lee JH, Ki HS, Yoon KW, Cho SB, Lee WS, Joo YE, Kim HS, Choi SK, Rew JS. [The trend of eradication rate of Helicobacter pylori infection and clinical factors that affect the eradication of first-line therapy]. Korean J Gastroenterol. 2010 Jun;55(6):368-75. doi: 10.4166/kjg.2010.55.6.368. Korean. PMID 20571304
- [Result] Bang SY, Han DS, Eun CS, Kim JE, Ahn SB, Sohn JH, Jeon YC, Kang JO. [Changing patterns of antibiotic resistance of Helicobacter pylori in patients with peptic ulcer disease]. Korean J Gastroenterol. 2007 Dec;50(6):356-62. Korean. PMID 18159172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: five hospitals affiliated with the Catholic University who visited from August 2011 to June 2012
Pre-assignment Details: Mutation test group ; Patients which are no detection of H. pyloriare were excluded
Groups:
- Convential AOM Group: The investigators do not perform mutation test in the conventional group apply metronidazole 500 mg tid, amoxicillin 1 g bid, rabeprazole 20 mg bid during 1 week
Period: Overall Study
Arm/Group | Conventional AOC Group | Mutation Test Group | Convential AOM Group
Started | 308 | 308 | 308
Completed | 282 | 193 | 277
Not Completed | 26 | 115 | 31
Not completed — Lost to Follow-up | 26 | 115 | 31

BASELINE CHARACTERISTICS:
Groups:
- Convential AOC Group: amoxicillin 1 g, bid , rabeprazole 20 mg bid, clarithromycin 500 mg bid during 1weeks
- Convential AOM Group: The investigators do not perform mutation test in the conventional group apply amoxicillin 1 g, bid , rabeprazole 20 mg bid, metronidazole 500mg tid during 1weeks
- Total: Total of all reporting groups
Arm/Group | Convential AOC Group | Mutation Test Group | Convential AOM Group | Total
Number analyzed (Participants) | 308 | 218 | 308 | 834
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 308 | 218 | 308 | 834
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (12.0) | 54.7 (12.2) | 56.2 (13.2) | 54.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 49 | 150 | 404
  Male | 103 | 169 | 158 | 430
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 308 | 218 | 308 | 834

OUTCOME MEASURES:

1. Primary Outcome: Helicobacter Pylori Eradication Rate
Description: Eradication was determined by the C13-urea breath test 6 to 8 weeks after the eradication therapy when PPIs had not been used for at least 2 weeks.
Time Frame: 8 weeks
Population: Each convential AOC, AOM group : 308 patients Mutation test gorup : H. pylori was not detected by PCR 90 patient , total 218 patient predicted prevalence - 50%, expected dropout rate -15%, predicted eradication rate - 80%, significance level - 0.05, statistical power - 90%
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Convential AOC Group | Mutation Test Group | Convential AOM Group
Number analyzed (Participants) | 308 | 218 | 308
percentage of participants | 75.9 [70.2 to 81.6] | 91.2 [88.9 to 93.4] | 79.1 [73.7 to 84.5]

ADVERSE EVENTS:
Arm/Group | Convential AOC Group | Convential AOM Group | Mutation Test Group
Serious Adverse Events (participants affected / at risk) | 0/308 | 0/308 | 0/218
Other Adverse Events (participants affected / at risk) | 0/308 | 0/308 | 0/218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes